CLINICAL TRIAL: NCT04974320
Title: Applying Novel Biomarkers to Identify MINOCA Rapidly and the Prognostic Value of Novel Biomarkers Among Patients With Acute Chest Pain: a Clinical Study
Brief Title: Rapid Identification of MINOCA Based on Novel Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Jiali Wang, deputy chief physician, Qilu Hospital of Shandong University
Other Study IDs: MINOCA QiluH
Record Dates: First submitted 2021-07-12; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Myocardial Infarction With Non-obstructive Coronary Arteries; Grow Stimulation Expressed Gene 2; Copeptin; Identification; Prognosis
MeSH Terms: conditions — MINOCA; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- MINOCA: All patients diagnosed with MINOCA in precision cohort (NCT04044066) will be included.
  Interventions: Biological: blood biomarkers
- acute myocardial infarction (AMI）: All patients diagnosed with acute myocardial infarction（AMI）in precision cohort (NCT04044066) will be included.
  Interventions: Biological: blood biomarkers
- unstable angina (UA): The patients diagnosed with unstable angina（UA) in precision cohort (NCT04044066) will be selected according to the matching method.
  Interventions: Biological: blood biomarkers
- MINOCA （multi-center）: The patients diagnosed with MINOCA in multi-center cohort will be included.
  Interventions: Biological: blood biomarkers

INTERVENTIONS:
Biological: blood biomarkers — All patients were obtained blood biomarkers: troponin, ST2, copeptin

SUMMARY:
Among the patients diagnosed as acute myocardial infarction by coronary angiography, 5%-25% of the patients did not find coronary artery obstructive lesions. These patients do not need PCI. The discovery and verification of clinical protocols for accurate identification of myocardial infarction in the absence of obstructive coronary artery disease（MINOCA）is a major issue that needs to be addressed.Novel biomarkers like grow stimulation expressed gene 2（ST2）can indicate the degree of coronary artery obstruction, copeptin is a biomarker of cardiac emergency state. No clinical studies have been conducted to evaluate whether the novel biomarkers combination regimen can diagnose or exclude MINOCA.

Our research aims to establish and validate a model for the recognition of MINOCA based on novel biomarkers (ST2, copeptin) and to evaluate the prognostic value of novel biomarkers among patients with acute chest pain.

DETAILED DESCRIPTION:
A cross-sectional study design will be used to evaluate the correlation between baseline novel biomarkers（ST2 and copeptin）and MINOCA, and to establish a discriminant model for the identification of MINOCA, and to verify its discriminant efficacy. A cohort study design will be used to evaluate the prognostic role of novel biomarkers in patients with acute chest pain.

On the basis of precision cohort (BIPASS), the project team will adopt the method of cross-sectional diagnostic experimental study design. ①Blood samples of MINOCA and AMI were extracted. According to the new biomarkers（ST2 and copeptin）reported in literature, the team will detect and combine them with troponin, and correct the covariate. And then establish the multivariate joint discriminant model. ②At the same time, according to the propensity score, patients will be selected from UA in a 1:1 matching ratio for modeling. The discriminant model for rapid recognition of MINOCA will be verified by internal cross validation and external validation. Based on this discriminant model, whether the combined application of three biomarkers in MINOCA diagnosis is superior to that of a single biomarker will also be evaluated. Patients with acute chest pain from multi-center will be selected to verify the accuracy of the rapid discriminant model of MINOCA applied to patients with acute chest pain.

ELIGIBILITY:
Inclusion Criteria:

* The clear diagnosis of MINOCA, acute myocardial infarction（AMI) and unstable angina（UA) in BIpass
* The clear diagnosis of MINOCA from the multi-center cohort

Exclusion Criteria:

* Prior surgery (cardiac or non-cardiac), trauma or clinically evident coagulopathic bleeding (e.g. gastrointestinal, genitourinary, et al)
* Patient with non-cardiac co-morbidities with life expectancy less than 12 months
* Patients unwilling or unable to comply with all clinical follow-up schedules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with MINOCA and acute myocardial infarction（AMI）in BIpass that meet the inclusion and exclusion criteria of this project will be included, and patients with unstable angina（UA）in BIpass that meet the inclusion and exclusion criteria of this project will be selected according to the matching method. This project will include multi-center MINOCA patients for external validation of the model.
Sampling Method: Non-Probability Sample
Enrollment: 2616 (Estimated)
Dates: Start 2021-06-05 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
MINOCA | 12 months
  The diagnosis of MINOCA is made immediately upon coronary angiography in a patient presenting with features consistent with an AMI, as detailed by the following criteria: universal AMI criteria; non-obstructive coronary arteries on angiography, defined as no coronary artery stenosis ⩾50% in any potential IRA; no clinically overt specific cause for the acute presentation.

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 12 months
  a composite of all-cause death, cardiac death, non-cardiac death, myocardial infarction or stroke

CONTACTS AND LOCATIONS:
Overall Officials: Jiali Wang, PhD,MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided